CLINICAL TRIAL: NCT00899821
Title: Head And Neck Cancer Immunotherapy Using Biodegradable Microspheres
Brief Title: Microsphere-Delivered Cytokines in Increasing Tumor Response in Lymphocytes From Patients With Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000280490; NYU-9916
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2008-12

CONDITIONS: Head and Neck Cancer
Keywords: recurrent metastatic squamous neck cancer with occult primary; untreated metastatic squamous neck cancer with occult primary; stage I squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the larynx; stage I squamous cell carcinoma of the lip and oral cavity; stage I squamous cell carcinoma of the nasopharynx; stage I squamous cell carcinoma of the oropharynx; stage I squamous cell carcinoma of the paranasal sinus and nasal cavity; stage II squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the larynx; stage II squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the nasopharynx; stage II squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent salivary gland cancer; salivary gland squamous cell carcinoma; stage I salivary gland cancer; stage II salivary gland cancer; stage III salivary gland cancer; stage IV salivary gland cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Salivary Gland Neoplasms | interventions — aldesleukin; Interleukin-12 Subunit p35; sargramostim; Immunologic Techniques; Biopsy

INTERVENTIONS:
Biological: aldesleukin
Biological: recombinant interleukin-12
Biological: sargramostim
Other: immunologic technique
Procedure: biopsy

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about how interleukin-2, interleukin-12, and GM-CSF delivered in microspheres increase the body's ability to kill tumor cells.

PURPOSE: This laboratory study is looking at microsphere-delivered cytokines to see if they increase tumor response in lymphocytes from patients with head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether local sustained delivery of cytokines (interleukin-2, interleukin-12, or sargramostim [GM-CSF]) in biodegradable microspheres augments antitumor response in human peripheral blood lymphocytes (PBLs) obtained from patients with squamous cell carcinoma of the head and neck, as evaluated in a human/SCID chimeric mouse model.
* Assess the potential of cytokine-loaded microspheres combined with dendritic cells (pulsed with tumor peptide) obtained from these patients to enhance long-term immunity against the tumor, as evaluated in a human/SCID chimeric mouse model.
* Evaluate the antitumor effect of the more effective approach (objective I or II) against established tumors in the mouse model.

OUTLINE: Biopsies of tumor are obtained during surgical resection. Patients undergo phlebotomy or leukapheresis to obtain peripheral blood lymphocytes (PBLs). PBLs, tumor tissue, and cytokine-loaded microspheres are coengrafted into SCID mice. Tumor growth and immune response are determined.

Dendritic cells are obtained from PBLs, expanded in culture, and pulsed with either autologous tumor cell lysates or peptide eluted from the tumor cells. The dendritic cells are coengrafted with tumor cells, PBLs, and cytokine-loaded microspheres into SCID mice. The mice are then challenged with autologous tumor cells, and antitumor response is determined.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma of the head and neck
* Tumor tissue shows engraftment in severe combined immunodeficient (SCID) mice or growth in tissue culture

PATIENT CHARACTERISTICS:

Age

* 20 to 80

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No known immunocompromised disease or condition
* No social, physical, or psychiatric condition that would preclude leukapheresis

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No concurrent immunosuppressive medication

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-06; Primary Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Local and sustained cytokine combinations in evaluating antitumor response in human peripheral blood lymphocytes obtained from patients with squamous cell carcinoma of the head and neck
Vaccine potential in provoking or enhancing long-term systemic immunity against head and neck cancer
Response rate

CONTACTS AND LOCATIONS:
Overall Officials: Moni A. Kuriakose, MD, Study Chair — NYU Langone Health